CLINICAL TRIAL: NCT07099495
Title: Reduced Functionality and Kinesiophobia in Patients With Heart Failure: Use of Neuromuscular Electrical Stimulation as an Alternative Therapeutic Strategy
Brief Title: REDUCED FUNCTIONALITY AND KINESIOPHOBIA IN PATIENTS WITH HEART FAILURE: USE OF ALTERNATIVE THERAPEUTIC STRATEGIES
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal do Rio Grande do Norte (Other)
Responsible Party: Principal Investigator, Patri-cia Angelica de Miranda Silva Nogueira, Principal Investigator, Universidade Federal do Rio Grande do Norte
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 84724024.6.0000.5537
Record Dates: First submitted 2025-07-07; First posted 2025-08-01 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Heart Failure; Heart Failure NYHA Class III; Heart Failure NYHA Class IV; Neuromuscular Electrical Stimulation (NMES); Kinesiophobia
Keywords: heart failure; neuromuscular electrical stimulation; kinesiophobia
MeSH Terms: conditions — Heart Failure; Kinesiophobia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Low Frequency Neuromuscular Electrical Stimulation (Active Comparator): Participants in this group will undergo low-frequency neuromuscular electrostimulation interventions, in accordance with the adopted intervention protocol, with assessments before, after, and at the end of the protocol to observe its effects.
  Interventions: Device: Low Frequency Neuromuscular Electrical Stimulation
- Medium Frequency Neuromuscular Electrical Stimulation (Active Comparator): Participants in this group will undergo medium-frequency neuromuscular electrostimulation interventions, in accordance with the adopted intervention protocol, with assessments before, after, and at the end of the protocol to observe its effects.
  Interventions: Device: Medium Frequency Neuromuscular Electrical Stimulation
- Neuromuscular Electrical Stimulation without generating contractility (Placebo Comparator): Participants in this group will undergo neuromuscular electrostimulation interventions at a frequency below the contractility threshold, comprising the placebo group, in accordance with the intervention protocol adopted, with assessments before, after, and at the end of the protocol to observe its effects.
  Interventions: Device: Neuromuscular Electrical Stimulation without generating contractility

INTERVENTIONS:
Device: Low Frequency Neuromuscular Electrical Stimulation — The surface electrodes will be placed on the upper lateral side of the quadriceps, 5 cm below the inguinal fold and 3 cm above the upper edge of the patella of both lower extremities, bilaterally and with a slight flexion of the knees. They will be fixed with bandages or tape, and conductive gel will be used below the electrodes. Each electrically stimulated contraction will have a frequency of 10 Hz, duration of 10 seconds (ON time: 10s), interspersed with a 20-second rest period (OFF time: 20s), with a pulse width of 400 µs. The protocol will last a total of 8 weeks, being performed 3 times a week, with application of the equipment for 30 minutes each day.
  Arms: Low Frequency Neuromuscular Electrical Stimulation
Device: Medium Frequency Neuromuscular Electrical Stimulation — The surface electrodes will be placed on the upper lateral side of the quadriceps, 5 cm below the inguinal fold and 3 cm above the upper edge of the patella of both lower extremities, bilaterally and with a slight flexion of the knees. They will be fixed with bandages or adhesive tape, and conductive gel will be used below the electrodes. Each electrically stimulated contraction will have a frequency of 50 Hz, duration of 10 seconds (ON time: 10s), interspersed by a period of 20 seconds of rest (OFF time: 20s), with a pulse width of 400 µs. The protocol will last a total of 8 weeks, being performed 3 times a week, with application of the equipment for 30 minutes each day.
  Arms: Medium Frequency Neuromuscular Electrical Stimulation
Device: Neuromuscular Electrical Stimulation without generating contractility — The surface electrodes will be placed on the upper lateral side of the quadriceps, 5 cm below the inguinal fold and 3 cm above the upper edge of the patella of both lower extremities, bilaterally and with a slight flexion of the knees. They will be fixed with bandages or adhesive tape, and conductive gel will be used below the electrodes. No muscle contractions will be generated. The protocol will last a total of 8 weeks, being performed 3 times a week, with application of the equipment for 30 minutes each day.
  Arms: Neuromuscular Electrical Stimulation without generating contractility

SUMMARY:
Introduction: Heart failure (HF) is a clinical syndrome that has advanced on a large scale concomitant with population aging and other factors. Thus, the search for alternatives that minimize the losses resulting from its structural and functional damage are important to optimize its treatments, with the primary objective of enabling the participation of these individuals in the most diverse daily tasks. Low-frequency (LF) or medium-frequency (MF) neuromuscular electrical stimulation (NMES) can be considered a resource to enable the improvement of vital and functional parameters of the population with HF intolerant to physical exercise, and it is also important to identify within these modalities which is most effective. In addition to these factors, kinesiophobia can be found in this population, and NMES can also be adopted as a strategy for kinesiophobia in these patients, with the objective of enabling the progression of behaviors. Objective: To evaluate and compare the effectiveness of LF and MF NMES on the indices of kinesiophobia and functionality in patients with HF. Methods: The research will be divided into two types of study: a double-blind randomized clinical trial (RCT) to evaluate NMES protocols, and a qualitative study with subsequent development and validation of a questionnaire to measure kinesiophobia in individuals with HF. The population included in the RCT will have their assessments (personal, socioeconomic, demographic data, Sit-to-Stand Test, kinesiological ultrasound and surface electromyography of the quadriceps muscles) conducted before their discharge from Hospital Nova Esperança (HNE), and after completion of the protocols at the same institution, in the city of João Pessoa - Paraíba. The application of NMES protocols will be carried out in the home environment (30 min/day, 3 times a week, for a total of 8 consecutive weeks). The population for the qualitative study and for the development of the questionnaire will consist of individuals diagnosed with HF of any etiology, compensated and able to perform kinesiotherapy activities, admitted to the HNE wards, between 24-48 hours before hospital discharge. An in-depth semi-structured interview will be conducted with these individuals, followed by the application of questionnaires developed based on the interviews, and the entire study will be conducted while the patients are hospitalized. Expected results: Regarding the first study, it is expected that patients treated with NMES will show improvements in clinical and functional variables, and these improvements may be more pronounced depending on the frequency applied. On the other hand, the qualitative study may reveal whether patients have fear of movement, even if they are clinically stable. The developed questionnaire will be well understood and have adequate psychometric qualities. Finally, it is expected that this knowledge can serve as a basis for optimizing the care of this patient population.

DETAILED DESCRIPTION:
Study 1 (double-blind randomized clinical trial) will be developed by recruiting individuals with chronic HF NYHA III-IV at the Hospital Nova Esperança (HNE), in the city of João Pessoa, state of Paraíba, Brazil, through advertising at the hospital where the participants' assessments will be performed (including patients who meet the study's eligibility criteria after hospital discharge). These individuals will be invited to participate in the study and instructed on its due procedures. To ensure the safety of the participants and reliability of the data, the medical records will be checked beforehand to ensure the necessary criteria are met. The researchers who will contribute to the study will be trained to perform the assessment of the participants, as well as to apply the LF and MF NMES protocol. The training will be offered by qualified professionals and the sequence and method of conducting the assessment and the NMES protocol will be recorded for the researchers involved. Strategies will be developed in advance to better organize the days, times, and logistics that seek to facilitate and optimize the conduct of the research, and will be planned according to the specificities of each researcher. Potential participants will be identified at the HNE together with the professionals of the service, who will maintain constant attention to identify patients who are eligible after their discharge. Once identified, they will contact the researchers to inform them, and the researcher responsible for this demand will go to the patient to provide explanations about the research, evaluate them, and ask for their telephone number to contact them after discharge. Other forms of recruitment will occur through active search in the aforementioned establishments and on social media. Randomization will be through the website randomization.com by a researcher who will not inform the evaluators, intervention researchers, or even the researcher who will perform the statistical analysis, about the groups in which these participants are located, leaving them blind. During randomization, participants will be allocated to three distinct groups: Intervention Group 1 (IG1): LF NMES protocol; Intervention Group 2 (IG2): MF NMES protocol; and Control Group (CG): NMES protocol without generation of muscle contractility. Four evaluators will participate in the study: researcher 1 will be responsible only for the evaluations, researchers 2 and 3 for the home application of the NMES protocols, and researcher 4 for randomization. The study will be double-blind, since researcher 1 and the participants will not be aware of the allocation of the subjects into the groups or the effects of the intervention. After the groups are formed, the research participants will be invited to come to the HNE outpatient clinic to perform the first day of evaluation before the start of the protocol. The evaluator will be a properly trained researcher who is blind to the intervention allocation group. This evaluation will include: personal, socioeconomic, and demographic data; collection of clinical data (history of the disease, ECHO results, and medications in use); vital signs (HR, RR, SpO2, and BP); lung, diaphragmatic, and quadriceps muscle ultrasound; lower limb perimeter; EMS of quadriceps muscles; 6MWT; application of the Lawton Scale and the Minnesota Living with Cardiac Insufficiency Questionnaire. After the day of the first assessment, the application of the GI1, GI2 and GC protocols will begin, which will occur for a total period of 8 weeks, 3 times/week, for 30 minutes on each day of application. The application days will be staggered, with a rest period between the scheduled days. The days and times will be assigned according to the availability of the participant and the researcher in charge. After 4 weeks of application of the protocol, they will return to the HNE outpatient clinic for a reassessment, which will have a specific day only for this purpose. After the reassessment, the application of the protocol will return. At the end of the 8 weeks, another reassessment will be performed, with the entire process being completed after 1 month of application of the protocol, with a follow-up.

In research number 2, for the process of constructing and validating the questionnaire, studies with different methodological designs will be carried out in two consecutive stages. The first stage will begin with the identification of the items that will make up the questionnaire. These items will be identified from a qualitative study with patients eligible for the research, through a semi-structured interview (which will be recorded for later analysis). The interview will be conducted with a guide of open-ended questions (between 3-5 questions) about the perceptions and/or concrete experiences of patients regarding their possible capabilities, fears or fear of performing physical activity. Participants will be recruited during their hospitalization, and their participation in the research will also occur during this same period. Immediately after this stage, the questionnaire items will be constructed, based on the main perceptions identified in the qualitative study and in the process of discussion and consensus of the researchers involved. The format of the questions and answers of the questionnaire will be defined after analysis of the qualitative data. Once the first version of the questionnaire is finalized, it will undergo a pre-test to assess the understanding of the items by the volunteers and health professionals of the service. Everyone will report their perception regarding the understanding and relevance of the questions. An item will undergo reformulation if less than 80% of those evaluated classify the term as incomprehensible or inadequate. The second stage, which corresponds to The validation of the questionnaire will also be performed with patients diagnosed with HF admitted to the service. The questionnaire will be given to the patients by the researcher, who will explain its purpose. Participants will have two days to return the completed questionnaire, to avoid recall bias. The informed consent form must be signed in duplicate by all participants. The test-retest reliability will be assessed by completing the questionnaire again, three days after the first, in a small sample of participants, approximately 30 subjects. Subsequently, the questionnaire will be applied to a representative sample of the hospital population to analyze its convergent and divergent validity, comparing it with other instruments and/or functional tests, such as the Anxiety and Depression Scale (HADS), Quality of Life (Minnesota Living with Cardiac Insufficiency), Exercise Tolerance (TSL1) and Surface Electromyography. Finally, clinical data will be extracted from the participants' medical records, as well as their length of hospital stay and the total period of care provided by the on-call physiotherapist to the participant being evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Individuals of both sexes;
* Age ≥ 18 years;
* Diagnosis of chronic HF;
* Symptoms compatible with Functional Class (FC) III-IV of the New York Heart Association (NYHA);
* Stable condition on pharmacological therapy;
* Absence of Acute Myocardial Infarction in the last three months prior to participant recruitment;
* Absence of an automatic internal cardioverter defibrillator (ICD) or cardiac pacemaker;

Exclusion Criteria:

* Individuals with hemodynamic instability, unstable angina, acute myocardial infarction during the period of application of the protocol and diagnosis of hypertrophic cardiomyopathy during the period of application of the protocol;
* Individuals with recent muscle or tendon injuries, muscular dystrophies, myopathies, unstable fractures, infections or deep vein thrombosis (DVT);
* Chronic need for oxygen therapy;
* Absence in reassessments;
* Refusal to participate in the research after its beginning.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2025-08-18 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Muscle strength | In the initial assessment, four weeks after the start of the intervention, at the end of the intervention (eight weeks of intervention), and one month after the complete conclusion of the protocol.
  A surface electromyograph (Miotool 400 - Miotec Equipamentos Biomédicos Ltda, POA, Brasil®) will be used to assess muscle production, strength and activation, calculating the maximum power that the patient will make in a voluntary isometric contraction of the quadriceps muscles (rectus femoris, vastus medialis and vastus lateralis), before and after the total NMES protocol.
Muscle thickness | At baseline, four weeks after the start of the intervention, at the end of the intervention (eight weeks of intervention), and one month after the complete conclusion of the protocol.
  Functional Kinesiological USG of the quadriceps muscles will be used to assess muscle thickness before starting the protocol, after 4 weeks and after the total intervention protocol with NMES, which may generate functional correlations with the protocol used. The evaluation protocol adopted will be that of Capmbell et al (1995) where quadriceps muscle thickness (QMT) will be quantified by a portable Mindray ultrasound, in B mode, in the supine position, with knees extended and relaxed.
Functional Capacity - 1-Minute Sit-to-Stand Test | At baseline, four weeks after the start of the intervention, at the end of the intervention (eight full weeks of intervention), and one month after the complete conclusion of the protocol.
  The individual is asked to sit and stand up in a standard-height chair (46-48 centimeters) positioned against a wall. The knees and hips should be flexed at 90 degrees, and the feet should be flat on the floor and hip-width apart. The patient's hands should rest on their hips and no support should be used. Over the course of one minute, the patient should sit and stand up from the chair repeatedly, aiming for as many times as possible. The test begins after a verbal command, and the patient will be notified when 15 seconds remain. The number of repetitions performed is counted and the modified Borg scale will be used to assess dyspnea and fatigue during and at the end of the test (BOHANNON & CROUCH, 2018).

SECONDARY OUTCOMES:
Participation in activities of daily living | At baseline, four weeks after the start of the intervention, at the end of the intervention (eight full weeks of intervention), and one month after the complete conclusion of the protocol.
  To assess the level of functional independence of research participants before, during and after the application of the protocol, the Lawton Scale will be used in the version translated and validated for the Portuguese language, which is a widely used instrument to assess individuals' participation in IADLs. The instrument consists of 7 items, each divided into three subitems, the main items being: telephone, travel, shopping, meal preparation, housework, medications and money. All items have three subitems, providing examples of specificities about the functional independence that the individual has when dealing with the points mentioned. The score ranges from 7 to 21.
Quality of life of individuals with Heart Failure | At baseline, four weeks after the start of the intervention, at the end of the intervention (eight full weeks of intervention), and one month after the complete conclusion of the protocol.
  The Minnesota Living with Cardiac Insufficiency Questionnaire, translated and validated in Portuguese, will be used to assess QoL before, after 4 weeks of application of the protocol, after full application, and 1 month later by follow-up of NMES, with 21 objective questions that assess physical, emotional and socioeconomic conditions. It offers a scale ranging from 0 to 5, with a final score ranging from 0 to 10, where higher scores are associated with worse QoL.

CONTACTS AND LOCATIONS:
Overall Officials: Patrícia A de Miranda Silva Nogueira, Doctorate degree (PhD), Study Director — Universidade Federal do Rio Grande do Norte
Locations (1):
- Av Capitão José Pessoa, 870, Jaguaribe, João Pessoa, Paraíba, Brazil

IPD SHARING:
Plan to Share IPD: Yes
All IPD that support the results of a publication will be shared.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: For the journal candidate for publication, from the transitional publication period, if necessary.
Access Criteria: They will be available to the journal applying for publication of the article, if necessary, to ensure the reliability of the study, by email or contact indicated by the journal.